CLINICAL TRIAL: NCT07306624
Title: A Multicenter, Phase 2 Clinical Trial Based on an Adaptive Design to Evaluate the Safety and Efficacy of Nelmastobart in Combination With Docetaxel in Patients With Advanced/Metastatic Non-Small Cell Lung Cancer Who Are Resistant or Intolerant to Platinum-based Chemotherapy and/or Immunotherapy
Brief Title: Nelmastobart in Combination With Docetaxel in Non Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: STCube, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STCUBE-004
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: BTN1A1; nsclc; immune check point inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nelmastobart 800mg+Docetaxel 75mg/m2 (Experimental): Nelmastobart 800mg+Docetaxel 75mg/m2 fixed
  Interventions: Drug: Nelmastobart and Docetaxel

INTERVENTIONS:
Drug: Nelmastobart and Docetaxel — Nelmastobart 800mg and Docetaxel 75mg/m2

SUMMARY:
A Multicenter, Phase 2 Clinical Trial Based on an Adaptive Design to Evaluate the Safety and Efficacy of Nelmastobart in Combination with Docetaxel in Patients with Advanced/Metastatic Non-Small Cell Lung Cancer Who Are Resistant or Intolerant to Platinum-based Chemotherapy and/or Immunotherapy

DETAILED DESCRIPTION:
This is a singble arm, open label, phase 2 study to evaluate safety and preliminary efficacy for Nelmastobart 800mg and docetaxel 75mg/m2 combination regimen for both AGA negative and positive NSCLC patients who have failed at least 1 line of treatment including platinum based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIb, IIIc, or IV 4 recurrent non-squamous NSCLC
* BTN1A1 TPS score ≥50
* Subjects with positive AGA must have progressed after At least 1 platinum-based chemotherapy and/or immunotherapy AND at least 1 locally approved targeted therapy appropriate to the AGA
* Subjects with negative AGA must have progressed after prior PD1/ (PDL therapy and/or platinum-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0- 1.
* Adequate organ function as described in the protocol
* Adequate cardiac function as described in the protocol
* For female or male patients with reproductive potential: Agree to use contraception throughout the study and at least 5 months after the last dose.
* Life expectancy of at least 3 months
* Has agreed to provide archival tissue

Exclusion Criteria:

* Known hypersensitivity to the active ingredients or excipients of the study drug.
* History of using Docetaxel for palliative therapy.
* Prior treatment with Cytotoxic chemotherapy or oral targeted therapy within 14 days.
* Investigational drugs within 5 half-lives.
* Monoclonal antibodies or ADCs within 4 weeks.
* Use or expected use of strong CYP3A4 inhibitors (e.g., ketoconazole) within 14 days prior to the first dose.
* Uncontrolled severe infection requiring IV treatment, or suspected infectious complications/fever.
* Requirement for continuous high-dose steroids (>10 mg/day prednisone equivalent) or immunosuppressants within 7 days (excluding Docetaxel premedication; intermittent/replacement therapies allowed).
* Pregnant or breastfeeding women.
* History of autoimmune disease requiring systemic treatment within the last 2 years
* Known active symptomatic or radiologically unstable CNS lesions
* History of stroke, unstable angina, MI, or NYHA Class III-IV symptoms within 6 months, or current Class II.
* Systolic BP 160 mmHg or Diastolic BP 100 mmHg, or hypertensive encephalopathy.
* History of ILD, organizing/drug-induced pneumonia, or active pneumonia on screening (mild asymptomatic fibrosis requires consultation).
* Recipients of allogeneic stem cell or solid organ transplants.
* Vaccination with live or attenuated live vaccines within 30 days.
* Maligancies other than NSCLC
* Failure to recover from prior anti-cancer therapy side effects to CTCAE Grade 1
* Wide-field bone marrow radiation (>30%) within 4 weeks, or limited palliative radiation within 2 weeks.
* Major surgery within 4 weeks or incomplete recovery from surgical side effects.
* Evidence of active HBV, HCV, or HIV infection (carriers with negative viral loads/RNA may be eligible).
* Clinically unstable pleural or peritoneal effusion (stable cases after intervention are allowed).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival by central reviewer | up to 3 years
  Time from first dose until the date of objective disease progression or death assessed by central reviewer

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  Time from first dose of study drug until the date of death
Progression Free Survival assessed by Investigator | Up to 3 years
  Time from first dose until the date of objective disease progression or death
Objective response rate, ORR | Up to 3 years
  Proportional of subjects with confirmed PR/CR, assessed by investigator and central reviewer
Disease control rate, DCR | Up to 3 years
  Proportion of subjects with confirmed CR, PR, and SD assessed by investigator and central reviewer based on RECIST v1.1
Duration of Response | Up to 3 years
  Time from the date of first objective response (CR or PR) after investigational drug administration to the first documented disease progression (PD) or death from any cause, with documentation of disease progression status and cause of death, assessed by investigator and central reviewer based on RECIST v1.1
Progression free survival rate | 6 month
  the proportion of patients without documented progression and alive 6 months after the first dose of study drug
Cmax | 3 weeks
  Maximum plasma concentration
Area under concentration-time curve | 15 weeks
  Area under the concentration-time curve during steady state
Adverse event | time from the date of the first dose of study drug until 30 days after last dose
  Incidence and severity of AE determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0

OTHER OUTCOMES:
Quality of life measured by EQ-5D-5L | until the end of treatment (Up to 3 years)
  Change from Baseline in Patient Reported Outcome EQ-5D-5L at Treatment Cycle 2 and beyond

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - The Catholic University of Korea St. Vincent's Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No